CLINICAL TRIAL: NCT00002116
Title: A Phase I/II Study of the Safety and Efficacy of Topical 1-(S)-(3-Hydroxy-2-Phosphonylmethoxypropyl)Cytosine Dihydrate (Cidofovir; HPMPC) in the Treatment of Refractory Mucocutaneous Herpes Simplex Disease in Patients With AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 218A; GS-93-301
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-12

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Herpes Simplex; Acquired Immunodeficiency Syndrome; Antiviral Agents; cidofovir
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Cidofovir

INTERVENTIONS:
Drug: Cidofovir

SUMMARY:
To evaluate the safety and tolerance of topical cidofovir (HPMPC) therapy for refractory mucocutaneous herpes simplex virus disease in AIDS patients. To determine whether topical HPMPC therapy can induce re-epithelialization and healing of refractory mucocutaneous herpes simplex virus disease in AIDS patients. To evaluate the virologic effects of topical HPMPC therapy on herpes simplex virus shedding from refractory lesions.

DETAILED DESCRIPTION:
Patients are randomized to receive topical therapy with placebo (vehicle alone) or HPMPC at either 0.3 or 1.0 percent once daily for 5 days. Patients are assessed to day 15; those with no significant toxicity are eligible to receive open-label topical HPMPC for up to 6 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy with AZT, ddI, ddC, or d4T.
* Oral trimethoprim/sulfamethoxazole.
* Dapsone.
* Atovaquone.
* Fluconazole.
* Rifabutin.
* Clarithromycin.

Patients must have:

* HIV seropositivity.
* Mucocutaneous herpes simplex virus (HSV) infection confirmed by previous viral culture and persisting without improvement despite at least 10 days of acyclovir at a minimum dose of 1 g/day (oral) or 15 mg/kg/day (intravenous).
* Measurable lesions.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Active medical problems sufficient to hinder study compliance or assessment of treatment effect.

Concurrent Medication:

Excluded:

* Acyclovir.
* Immunomodulators (such as corticosteroids or interferons).
* Lymphocyte replacement therapy.
* Biologic response modifiers.
* Ganciclovir.
* Foscarnet.
* Vidarabine.
* Topical trifluridine.
* Other investigational drugs (except d4T).
* Amphotericin.
* Intravenous therapy for PCP.
* Chemotherapeutic agents.

Prior Medication:

Excluded within 14 days prior to study entry:

* Immunomodulators (such as corticosteroids or interferons).
* Lymphocyte replacement therapy.
* Biologic response modifiers.
* Ganciclovir.
* Foscarnet.
* Vidarabine.
* Topical trifluridine.
* Other investigational drugs with potential anti-HSV activity.
* Amphotericin.
* Intravenous therapy for PCP.

Excluded within 4 weeks prior to study entry:

* Chemotherapeutic agents.

Required:

* At least 10 days of prior acyclovir at a minimum dose of 1 g/day (oral) or 15 mg/kg/day (intravenous).

Substance abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of North Carolina Hosps, Chapel Hill, North Carolina
  - Park Plaza Hosp, Houston, Texas
  - Univ of Washington / Viral Disease Clinic, Seattle, Washington
- Univ of British Columbia / Univ Hosp, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Acyclovir-resistant herpes: expanded access available for cidofovir gel (Forvade). AIDS Treat News. 1997 Feb 7;(No 264):5. PMID 11364104